CLINICAL TRIAL: NCT02430467
Title: Caregiver-Guided Pain Management Training in Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Palliative Care Research Cooperative Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00057512; 1R01NR015348-01 (NIH)
Record Dates: First submitted 2015-04-24; First posted 2015-04-30 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caregiver-guided pain management training protocol (CG-PMT) (Active Comparator): Patient-caregiver dyads in the CG-PM arm of the study will receive 3 50-minute sessions via Skype with a masters-level therapist over a 3-week period. The intervention integrates educational information about cancer pain and its management with a behavioral training program to teach patients and caregivers pain coping skills including relaxation, imagery, and activity pacing, and to teach caregivers how to guide and coach the patient in the practice and application of these pain control techniques
  Interventions: Behavioral: Caregiver-guided pain management training (CG-PMT)
- Enhanced treatment-as-usual (TAU) (Active Comparator): Patient-caregiver dyads in the Enhanced TAU condition will receive the same educational video and booklet on cancer pain and its management that is used as part of the CG-PMT intervention. They will also receive iPads with icons linked to reputable websites that provide educational information on cancer including cancer pain (e.g., ACS, NCI) and will be encouraged to utilize them for information and support. However, they will not meet with a study interventionist nor receive any training in behavioral pain coping skills.
  Interventions: Behavioral: Enhanced treatment-as-usual (TAU)

INTERVENTIONS:
Behavioral: Caregiver-guided pain management training (CG-PMT) — Patient-caregiver dyads in the CG-PM arm of the study will receive 3 50-minute sessions via Skype with a masters-level therapist over a 3-week period. The intervention integrates educational information about cancer pain and its management with a behavioral training program to teach patients and caregivers pain coping skills including relaxation, imagery, and activity pacing, and to teach caregivers how to guide and coach the patient in the practice and application of these pain control techniques.
  Arms: Caregiver-guided pain management training protocol (CG-PMT)
Behavioral: Enhanced treatment-as-usual (TAU) — Patient-caregiver dyads in the Enhanced TAU condition will receive the same educational video and booklet on cancer pain and its management that is used as part of the CG-PMT intervention. They will also receive iPads with icons linked to reputable websites that provide educational information on cancer including cancer pain (e.g., ACS, NCI) and will be encouraged to utilize them for information and support. However, they will not meet with a study interventionist nor receive any training in behavioral pain coping skills.
  Arms: Enhanced treatment-as-usual (TAU)

SUMMARY:
The purpose of this study is to develop more effective ways to help patients and their caregivers cope with cancer pain. The investigators are looking at the usefulness of a Caregiver-Guided Pain Management Training Intervention versus Pain Education.

DETAILED DESCRIPTION:
The primary aim of this study is to test the efficacy for the Caregiver-Guided Pain Management Training intervention to improve the caregiver's self-efficacy for helping the patient manage pain. Secondary aims include testing the effectiveness of the CG-PMT intervention to improve patient pain severity, patient self-efficacy for pain management and patient psychological distress, as well as short-term caregiver adjustment and caregiver adjustment following the patient's death.

In this multi-site study, 236 dyads (patients with cancer pain and their family caregivers) will be randomized to either a Caregiver-Guided Pain Management Training protocol or to an Enhanced Treatment-as-Usual control condition. Dyads in the Caregiver-Guided Pain Management condition will receive three one-hour sessions conducted via videoconference. Dyads in the Enhanced Treatment-as-Usual condition will receive educational material about cancer pain and its management but will not receive any study-related treatment sessions. Assessments will be conducted with patients and caregivers before and after treatment, and with caregivers 3 months and 6 months following the patient's death. The primary hypothesis to be tested is that caregivers who receive the intervention will report significantly higher levels of self-efficacy for helping the patient manage pain than caregivers in the control condition. Secondary aims will focus on (a) improvements in short-term caregiver adjustment as well as caregiver adjustment following the patient's death, and (b) patient pain severity, self-efficacy for pain management, and psychological distress.

ELIGIBILITY:
Patient Inclusion Criteria:

1. clinical diagnosis Stage 4 solid or hematologic malignancy and nonresectable Stage 3 gastrointestinal (GI) cancer
2. life expectancy of < 1 month
3. worst pain in the past 2 weeks greater than or equal to 4 on the 0-10 pain scale,
4. have an identified caregiver who is also willing to participate,
5. at least 18 years old, 6) fluent in English.

Caregiver Inclusion Criteria:

1. at least 18 years old
2. fluent in English

Patient Exclusion Criteria:

1. Palliative Performance Scale rating <40,
2. current external radiation therapy for reduction of pain
3. unable to provide informed consent or complete study procedures as determined by clinical or study staff.

Caregiver Exclusion Criteria:

1) unable to provide informed consent or complete study procedures as determined by clinical or study staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2015-07; Primary Completion 2018-11-01 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Change in caregiver self-efficacy for helping the patient manage pain | baseline, post-intervention (3 weeks)
  Caregiver Self-Efficacy Scale

SECONDARY OUTCOMES:
Change in caregiver strain | baseline, following intervention (3 weeks)
  Caregiver Strain Index
Change in caregiver satisfaction | baseline, following intervention (3 weeks)
  Caregiving Satisfaction Scale
Change in caregiver psychological distress | baseline, following intervention (3 weeks)
  Center for Epidemiology Studies Short Depression Scale
Change in caregiver psychological distress | following death of patient (3 mos & 6 mos)
  Trait Anxiety Scale
Change in caregiver health behaviors | following death of patient (3 mos & 6 mos)
  Self-Administered Comorbidity Questionnaire
Change in caregiver global health rating | following death of patient (3 mos & 6 mos)
  Global health rating
Change in patient pain | baseline, post-intervention (3 weeks)
  Brief Pain Inventory
Change in patient self-efficacy | baseline, post-intervention (3 weeks)
  Patient Self-Efficacy Scale
Change in patient psychological distress | baseline, post-intervention (3 weeks)
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Laura Porter, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Porter LS, Steel JL, Fairclough DL, LeBlanc TW, Bull J, Hanson LC, Fischer S, Keefe FJ. Caregiver-guided pain coping skills training for patients with advanced cancer: Results from a randomized clinical trial. Palliat Med. 2021 May;35(5):952-961. doi: 10.1177/02692163211004216. Epub 2021 Mar 29. PMID 33775175
- [Derived] Porter LS, Samsa G, Steel JL, Hanson LC, LeBlanc TW, Bull J, Fischer S, Keefe FJ. Caregiver-guided pain coping skills training for patients with advanced cancer: Background, design, and challenges for the CaringPals study. Clin Trials. 2019 Jun;16(3):263-272. doi: 10.1177/1740774519829695. Epub 2019 Feb 19. PMID 30782014